CLINICAL TRIAL: NCT00885807
Title: Psychometric Validation of the Weiss Functional Impairment Rating Scale and the Weiss Symptom Record in Patients With Attention-Deficit Hyperactivity Disorder
Brief Title: A Prospective Chart Review to Validate the WFIRS (Weiss Functional Impairment Rating Scale)
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Eli Lilly and Company (Industry); Purdue Pharma LP (Industry); Shire (Industry)
Responsible Party: Dr. Margaret Weiss, University of British Columbia
Other Study IDs: H05-70402
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: ADHD; WFIRS; WSR
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to evaluate the psychometric validation of the Weiss Functional Impairment Rating Scale and the Weiss Symptom Record. It is hypothesized that the Weiss Functional Impairment Rating Scale has strong psychometric properties and good convergent validity with other measures of functioning and discriminant validity from symptoms and quality of life.

DETAILED DESCRIPTION:
The measures for this rating scale were developed at the request of the Canadian Attention Deficit Disorder Resource Alliance to provide clinician friendly tools free of charge as a way of improving screening for ADHD and comorbidity.

Patients are consented during clinic visits and agree to allow use of clinic data for the purpose of this research. They complete additional measure(s) for the purpose of the study. The data is then entered.

Internal consistency will be measured using Cronbach's alpha. Convergent, concurrent and discriminant validity will be measured using Pearson correlations. Domain reliability is determined with factor analysis. Up to 220 patients will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Compliance to complete the WFIRS is key to inclusion.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People with ADHD from 7 years of age
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2006-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret D. Weiss, MD, Ph.D, Principal Investigator — University of British Columbia; Chistopher Gibbins, MD, Study Director — BC Children's & Women's Hospital, Vancouver; Grant Iverson, MD, Study Director — University of British Columbia; Brian Brooks, MD, Study Director — BC Children's & Women's Hospital, Vancouver; Li Ying Lu, MD, Study Director — BC Children's & Women's Hospital, Vancouver
Locations (1):
- Provincial ADHD Program, BC Children's & Women's Health Centre, Vancouver, British Columbia, Canada